CLINICAL TRIAL: NCT02335268
Title: Prospective Validation of a Predictive Model of Response to Romiplostim in Patients With IPSS Low or Intermediate-1 Risk Myelodysplastic Syndrome (MDS) and Thrombocytopenia - the EUROPE-trial
Brief Title: Validation of a Predictive Model of Response to Romiplostim in Patients With IPSS Low or Intermediate-1 Risk MDS and Thrombocytopenia
Acronym: EUROPE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gesellschaft fur Medizinische Innovation - Hamatologie und Onkologie mbH (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 440/47
Record Dates: First submitted 2015-01-07; First posted 2015-01-09 (Estimated); Results first posted 2023-07-14 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-07

CONDITIONS: Myelodysplastic Syndromes
Keywords: MDS classified as IPSS low/int-1
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — romiplostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Experimental): Stratification into group 1 if Score (Baseline-TPO Level and previous thrombocyte transfusions) are +3
  TPO based model to predict subsequent response to romiplostim in MDS patients with IPSS Low/Int-1 according to a model developed by Sekeres et. al./ BJH 2014
  Interventions: Drug: N-Plate / romiplostim
- Group 2 (Experimental): Stratification into group 2 if Score (Baseline-TPO Level and previous thrombocyte transfusions) are -1 or -2
  TPO based model to predict subsequent response to romiplostim in MDS patients with IPSS Low/Int-1 according to a model developed by Sekeres et. al./ BJH 2014
  Interventions: Drug: N-Plate / romiplostim
- Group 3 (Experimental): Stratification into group 3 if Score (Baseline-TPO Level and previous thrombocyte transfusions) are -6
  TPO based model to predict subsequent response to romiplostim in MDS patients with IPSS Low/Int-1 according to a model developed by Sekeres et. al./ BJH 2014
  Interventions: Drug: N-Plate / romiplostim

INTERVENTIONS:
Drug: N-Plate / romiplostim — medical intervention in 3 patient groups (MDS patients with IPSS Low/Int-1) that are stratified according to their baseline TPO-Level and previous transfusions

SUMMARY:
There are currently no licensed drugs in the EU to treat thrombocytopenia in MDS patients classified as IPSS low/int-1. Prior studies with romiplostim (a TPO receptor agonist) in MDS found that baseline concentration of TPO as well as transfusion history were predictive of subsequent response in a retrospective model. The current prospective study has the aim to explore whether both pretreatment variables (endogenous TPO, TPO-level, platelet transfusion history) can predict the response to subsequent short-term treatment with romiplostim.

DETAILED DESCRIPTION:
Myelodysplastic syndromes (MDS) are a heterogeneous group of hematologic malignancies of the pluripotent hematopoietic stem cells characterized by clonal hematopoiesis, progressive bone marrow failure, and the propensity to transform to acute myeloid leukemia (AML) (Malcovati et al., 2013).

There are currently no licensed drugs in the EU to treat thrombocytopenia in MDS patients classified as IPSS low/int-1. Prior studies with romiplostim (a TPO receptor agonist) in MDS found that baseline concentration of TPO as well as transfusion history were predictive of subsequent response in a retrospective model.

Classically, MDS is associated with apoptosis and excessive proliferation, resulting in a combination of a hyper-cellular marrow and peripheral cytopenia. The rationale for using romiplostim in MDS is to stimulate normal progenitor cells to increase platelet counts. Upon correction of thrombocytopenia, responding MDS patients should have a decreased risk of bleeding and a reduction in platelet transfusions (Giagounidis et al., 2014). This reduction in platelet transfusions may in turn decrease the risks of alloimmunization and the resultant morbidity and costs associated with that condition.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet the following inclusion/exclusion criteria to be eligible for the study.
* Must understand and voluntarily sign the informed consent form
* Age older 18 years at the time of signing the informed consent form
* Must be able to adhere to the study visit schedule and other protocol requirements
* Diagnosis of MDS using the 2008 WHO classification for myeloid neoplasms as assessed during the screening period
* Per MDS IPSS, low or intermediate-1 risk MDS as assessed during the screening period
* The mean of the 2 platelet counts taken within 4 weeks prior to stratification must be:
* ≤ 30 x 109/L (with no individual count > 30 x 109/L during the screening period), with or without a history of bleeding associated with the diagnosis of MDS, OR
* < 50 x 109/L (with no individual count >60 x 109/L during the screening period), with a history of bleeding associated with the diagnosis of MDS (A standard of care platelet count taken prior to Informed consent may be used as 1 of the 2 counts taken within 4 weeks prior to stratification)
* Adequate liver function, as evidenced by ALT ≤ 3 times the laboratory normal range, AST ≤ 3 times the laboratory normal range and total bilirubin ≤ 2 times the laboratory normal range
* Bone marrow aspirate (central diagnostics) with cytogenetics (local) within 8 weeks of starting first dose of investigational product
* Female subjects of childbearing potential† must:
* Agree to use, and be able to comply with, effective contraception without interruption, 4 weeks before starting study drug, throughout study drug therapy and for 4 weeks after the end of study drug therapy, even if she has amenorrhoea. This applies unless the subject commits to absolute and continued abstinence confirmed on a monthly basis. Male patients who wish to participate in the study and their partner may become pregnant must agree also to reliable contraception during the study and for three months thereafter.

The following are effective methods of contraception*

* Implant, - Levonorgestrel-releasing intrauterine system (IUS), Medroxyprogesterone acetate depot, Tubal sterilization, Sexual intercourse with a vasectomised male partner only; Ovulation inhibitory progesterone-only pills (i.e., desogestrel)
* Agree to have a medically supervised pregnancy test with a minimum sensitivity of 25 mIU/ml not more than 3 days before the start of study medication once the subject has been on effective contraception for at least 4 weeks. This requirement also applies to women of childbearing potential who practice complete and continued abstinence.

Exclusion Criteria:

* Pregnant or lactating females
* IPSS intermediate-2 or high-risk
* ≥ 5% blasts in the bone marrow as determined by central morphology during screening
* Previous treatment with any thrombopoietic growth factor
* Prior history of hematopoietic stem cell transplantation, leukemia, aplastic anemia or other non-MDS related bone marrow stem cell disorder
* Active or uncontrolled disease including infections or cancer
* Unstable angina, congestive heart failure (NYHA > class II), uncontrolled hypertension
* History of arterial thrombosis (e.g., stroke or transient ischemic attack) within the past year
* History of venous thrombosis that currently requires anti-coagulation therapy
* Prior use of sc or iv AZA.
* Receipt of G-CSF, peg-G-CSF, or GM-CSF,IL-11, ESA or LEN within 4 weeks of the first dose of romiplostim
* Planned receipt of peg-G-CSF or GM-CSF after the first dose of investigational product
* Subjects of reproductive potential who are not using adequate contraceptive precautions, in the judgment of the investigator. A double barrier method is defined as 2 methods of contraception, for example 2 actual barrier methods, or 1 actual barrier method and 1 hormonal method.
* Known hypersensitivity to any recombinant E. coli-derived product (eg, Nplate, Infergen, Neupogen, Somatropin, and Actimmune)
* Inability to comply with study procedures.
* Subject currently is enrolled in or has not yet completed at least 30 days since ending other investigational device or drug study(s)
* Any serious medical condition or psychiatric illness that will prevent the subject from signing the informed consent form or will place the subject at unacceptable risk if he/she participates in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2015-05-21 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Platzbecker, Prof. Dr., Study Director — University of Dresden; Lionel Ades, Prof. Dr., Study Director — Groupe Francophone des Myelodysplasies
Locations (36):
- France (22):
  - CH, Annecy
  - CH Victor Dupouy, Argenteuil
  - CH Henri Duffaut, Avignon
  - CHU de Haut Lévèque, Bordeaux
  - CHRU Côte de Nacre, Caen
  - CHU Estaing, Clermont-Ferrand
  - CHU, Grenoble
  - CH, Le Mans
  - CHRU, Limoges
  - CH Lyon sud, Lyon
  - IPC, Marseille
  - CH, Meaux
  - Clinique Beausoleil, Montpellier
  - CHU Brabois, Nancy
  - Centre Catherine de Sienne, Nantes
  - Polyclinique Le Languedoc, Narbonne
  - CHR, Orléans
  - Hôpital Cochin, Paris
  - Hôpital Saint Louis, Paris
  - CHU, Poitiers
  - Centre Henri Becquerel, Rouen
  - Hôpital Bretonneau, Tours
- Germany (14):
  - MVZ Onkologischer Schwerpunkt am Oskar-Helene-Heim, Berlin
  - Vivantes Klinikum am Urban / Hämatologie Onkologie, Berlin
  - Klinikum Chemnitz gGmbH / Klinik für Innere Medizin III, Chemnitz
  - Universitätsklinikum Dresden / Medizinische Klinik I, Dresden
  - Marienhospital Düsseldorf GmbH / Innere Medizin u. Hämatologie, Düsseldorf
  - Universitätsklinikum Halle (Saale) / Klinik für Innere Medizin IV, Halle
  - Universitätsklinikum Hamburg-Eppendorf /Onkologisches Zentrum, Hamburg
  - Medizinische Hochschule Hannover / Hämatologie u. Onkologie, Hanover
  - Universitätsklinikum Mannheim / Klinik III / Hämatologie, Onkologie, Mannheim
  - Klinikum Rechts der Isar, Tumortherapiezentrum, München
  - MVZ für Blut u. Krebserkrankungen, Potsdam
  - Universitätsklinikum Ulm / Klinik Innere Medizin III, Ulm
  - Onkologische Gemeinschaftspraxis, Weilheim
  - Rems-Murr-Kliniken Winnenden / Hämatologie, Onkologie, Winnenden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From May 2015 through July 2019, a total of 125 patients were screened at 19 study sites in France, 9 study sites in Germany and 1 study site in Czech Republic. Of them, 77 were eligible for study participation.
Pre-assignment Details: 77 patients were assigned into two different model groups at the time of screening based on previous platelet transfusion events (PTE) and centrally assessed TPO serum levels. 51 patients were assigned to Group A (TPO < 500 ng/L and PTE < 6 units/past year) and 26 patients to Group B+C (TPO > 500 ng/L, and/or PTE ≥ 6 units/past year).
Groups:
- Model Group A: Starting dose 750 µg of romiplostim once a week (7d ± 2d), subcutaneous injection, 4 months maximum duration for responders treatment period was extended for up to 1 year (8 months extension period). The dose was adjusted based on the subject's platelet count.
- Model Groups B+C: Starting dose 750 μg of romiplostim once a week (7d ± 2d), subcutaneous injection, 4 months maximum duration for non-responders. The dose was adjusted based on the subject's platelet count.
Period: Overall Study
Arm/Group | Model Group A | Model Groups B+C
Started | 51 | 26
Completed | 34 | 20
Not Completed | 17 | 6
Not completed — Physician Decision | 5 | 1
Not completed — Lack of Efficacy | 2 | 1
Not completed — Adverse Event | 5 | 2
Not completed — increase blasts | 2 | 0
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Model Group A | Model Groups B+C | Total
Number analyzed (Participants) | 51 | 26 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.6 (10.3) | 71.2 (8.3) | 72.1 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 10 | 28
  Male | 33 | 16 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 49 | 23 | 72
  Other | 2 | 3 | 5
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.46 (3.99) | 28.03 (4.44) | 26.97 (4.18)

OUTCOME MEASURES:

1. Primary Outcome: Hematologic Improvement of Platelets (HI-P) After 4 Months on Therapy
Description: The primary efficacy endpoint was the rate of HI-P defined as an absolute increase of platelet count to ≥ 30/nL for patients starting at > 20/nL or an increase of platelets from < 20/nL to > 20/nL and by at least 100%, according to IWG 2006 criteria lasting for ≥ 8 weeks after at least 16 Weeks of romiplostim treatment.
Time Frame: after 4 months on therapy (week 16)
Measure: Median (Full Range); unit: platelets (/nL)
Arm/Group | Model Group A | Model Groups B+C
Number analyzed (Participants) | 34 | 22
platelets (/nL) | 71.75 [-15.5 to 342.5] | 18.75 [-25.0 to 161.0]

2. Secondary Outcome: Cumulative Hematologic Improvement
Description: Cumulative rate of hematologic improvement of platelets (HI-P), erythrocytes (HI-E) and neutrophil granulocytes (HI-N).
  None of the patients achieved simultaneous response of HI-P, HI-E and HI-N.
Time Frame: week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Model Group A | Model Groups B+C
Number analyzed (Participants) | 51 | 26
Participants
  yes | 0 | 0
  no | 51 | 26

3. Secondary Outcome: The Incidence of Disease Progression to Higher Stage MDS or AML
Description: The incidence of disease progression to higher stage MDS or AML according to WHO (increase in blast percentage of ≥ 20 %)
Time Frame: week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Model Group A | Model Groups B+C
Number analyzed (Participants) | 51 | 26
Participants
  yes | 6 | 2
  no | 45 | 24

4. Secondary Outcome: Increase of Peripheral Blasts During Therapy
Time Frame: week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Model Group A | Model Groups B+C
Number analyzed (Participants) | 51 | 26
Participants
  < 5% | 31 | 15
  5%-10% | 0 | 0
  10%-20% | 0 | 0
  > 20% | 0 | 0
  missing | 20 | 11

5. Secondary Outcome: Association of the Presence of Certain Mutations With Disease Progression in a Retrospective Analysis
Time Frame: week 16
Measure: Count of Participants; unit: Participants
Groups:
- Full Analysis Set: The primary dataset for analysis is the full analysis set which is derived from all patients who fulfilled the inclusion criteria and gave their written informed consent.
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 77
Participants
  no | 69
  yes | 8

6. Secondary Outcome: Incidence of Bleeding Events
Time Frame: up to 12 months
Measure: Mean (Standard Deviation); unit: bleeding events per patient week
Arm/Group | Model Group A | Model Groups B+C
Number analyzed (Participants) | 51 | 24
bleeding events per patient week | 0.263 (0.476) | 0.249 (0.363)

7. Secondary Outcome: Type, Incidence and Severity of All Adverse Events Including Clinically Significant Changes in Laboratory Values
Time Frame: up to 12 months
Measure: Number; unit: events
Arm/Group | Model Group A | Model Groups B+C
Number analyzed (Participants) | 51 | 26
events | 499 | 159

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: Patients were asked to each visit whether they have experienced AEs or SAEs.
Arm/Group | Model Group A | Model Groups B+C
All-Cause Mortality (participants affected / at risk) | 0/51 | 1/26
Serious Adverse Events (participants affected / at risk) | 12/51 | 8/26
Other Adverse Events (participants affected / at risk) | 10/51 | 5/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Model Group A (N=51) | Model Groups B+C (N=26)
Hemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Central venous catheterization (Surgical and medical procedures) | 1 (1) | 0 (0)
AML (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Mucosal hemorrhage (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Testicular torsion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Drug-specific antibody (Investigations) | 1 (1) | 0 (0)
Monocyte count increased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Physical examination (Investigations) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal angiectasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis migration (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic mass (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Viral rash (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Model Group A (N=51) | Model Groups B+C (N=26)
Hematoma (Vascular disorders) | 4 (4) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Blast cells present (Investigations) | 5 (5) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 7 (7) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0)
Injection site hematoma (General disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/68/NCT02335268/Prot_SAP_000.pdf